CLINICAL TRIAL: NCT01296984
Title: A Registry Based Study of Clinical Results and of Health and Wellbeing in Patients After Abdominoperineal Resection for Rectal Cancer
Brief Title: Oncological and Functional Result of AbdominoPerineal Extra Levator Resection for Distal Rectal Cancer
Acronym: APER
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Swedish Cancer Foundation (Other)
Responsible Party: Principal Investigator, Eva Angenete, M.D., Ph.D., Sahlgrenska University Hospital
Other Study IDs: SSORG APER
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; APR
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Extralevator APR: The perineal part of the APR is done with the intent to create a cylindrically shaped specimen thus removing part of or the entire levator muscle with the specimen.
- Traditional APR: The perineal part of the APR is performed with the intent to remove the tumour with CRM free of tumour and the levator left in place.

SUMMARY:
The aim of the project is to evaluate the oncological and functional outcome of the more extensive perineal dissection - i.e the extra levator resection - in abdominoperineal resections in patients with rectal cancer.

Hypothesis: Extra levator perineal resection reduces local recurrence three year postoperatively compared to traditional abdominoperineal resection and improves QoL 2-4 years postoperatively.

DETAILED DESCRIPTION:
Low rectal cancer treated surgically by abdominoperineal resection (APR) has worse outcome than other rectal cancers operated with low anterior resection. In order to improve the outcome in the APR group a more extensive surgical procedure - the extra levator APR - has been suggested. This study aims to investigate both the oncological and the functional outcome of this method as compared to the traditional APR.

Method: All Swedish patients undergoing abdominoperineal resection for rectal cancer 2007-2009 will be analysed regarding operative technique (traditional or extra levator resection). Data on all patients regarding pre op TNM classification, pathological report and local recurrence will be collected from the Swedish Rectal Cancer registry. A validated QoL form will be sent to each patient to further investigate the functional outcome, health economy and Quality of Life 2-4 years postoperatively.

Data will be analysed regarding 3 year recurrence rate (primary endpoint) as well as functional result and QoL (secondary endpoints) in the two different groups - i.e traditional and extra levator APR.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer operated with APR 2007-2009

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All swedish patients registerd in the swedish rectalcancer registry undergoing APR 2007-2009
Sampling Method: Non-Probability Sample
Enrollment: 1319 (Actual)
Dates: Start 2011-02; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
3-year local recurrence | 3 years postoperatively
  Local recurrence of rectal cancer 3 years after APR

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  postoperative morbidity: wound infection, deep infections, other infections, wound necrosis, pain, pneumonia, thrombosis
Reoperation, readmittance and mortality | 12 months
  Re-operation/s, length of hospital stay/s, re-admittance/s, mortality all within 12 months of primary surgery
Late morbidity | 24-48 months postoperatively
  Late morbidity and functional disorders: prolonged wound healing, late infections, limping, pain, sitting problems, urinary incontinence, erectile dysfunction, stoma related dysfunction
Quality of Life | 24-48 months postoperatively
  Patient experienced health and QoL 24-48 months postoperatively
Health economy | 24-48 months postoperatively
  Health economy analysis of resource consumption
Stoma function | 24-36 months postop
  Assessment of stoma function related both to construction and surgical technique and patient position

CONTACTS AND LOCATIONS:
Locations (1):
- SSORG, Sahlgrenska Universitetssjukhuset, Område 2, Gothenburg, Västra Götalandsregionen, Sweden

REFERENCES:
- [Derived] Gonzalez E, Holm K, Wennstrom B, Haglind E, Angenete E. Self-reported wellbeing and body image after abdominoperineal excision for rectal cancer. Int J Colorectal Dis. 2016 Oct;31(10):1711-7. doi: 10.1007/s00384-016-2628-0. Epub 2016 Aug 10. PMID 27506432
- [Derived] Asplund D, Prytz M, Bock D, Haglind E, Angenete E. Persistent perineal morbidity is common following abdominoperineal excision for rectal cancer. Int J Colorectal Dis. 2015 Nov;30(11):1563-70. doi: 10.1007/s00384-015-2328-1. Epub 2015 Aug 6. PMID 26245948
- [Derived] Prytz M, Angenete E, Haglind E. Abdominoperineal extralevator resection. Dan Med J. 2012 Sep;59(9):A4366. PMID 22951192